CLINICAL TRIAL: NCT07116499
Title: A Phase IIa, Multicenter, Randomized, Double-Blind, Placebo-Controlled Crossover Study of K-645 in the Treatment of Multiple Migraine Attacks
Brief Title: A Study of K-645 in the Treatment of Multiple Migraine Attacks
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped for futility based on an interim analysis of efficacy.
Sponsor: Kallyope Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: K-645 P003
Record Dates: First submitted 2025-08-07; First posted 2025-08-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Acute Migraine

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, 3-period crossover study. In each period, participants will treat a single migraine attack. Participants will receive a different treatment in each of the three periods: placebo, K-645 dose level 1, or K-645 dose level 2.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study where the Sponsor, site staff and participants will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence 1 (Experimental)
  Interventions: Drug: Placebo; Drug: K-645 dose level 1; Drug: K-645 dose level 2
- Treatment Sequence 2 (Experimental)
  Interventions: Drug: Placebo; Drug: K-645 dose level 1; Drug: K-645 dose level 2

INTERVENTIONS:
Drug: Placebo — Single oral dose of matching placebo
Drug: K-645 dose level 1 — Single oral dose of K-645 dose level 1
Drug: K-645 dose level 2 — Single oral dose of K-645 dose level 2

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, 3-period crossover study to evaluate the safety, tolerability, and efficacy of two dose levels of K-645 in the treatment of patients with acute migraine.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Be a male or female, age 18 to 65 years, inclusive, at the time of signing informed consent.
2. Patient has greater than a one-year history of migraine with or without aura as defined by International Headache Society (IHS) criteria 1.1 and 1.2 and his/her migraines typically last between 4 to 72 hours, if untreated (refer to International Classification of Headache Disorders [ICHD] III Attachment for IHS migraine definitions) as documented in the patient's medical records from his/her treating physician and confirmed by the investigator.
3. Patient has had ≥2 and ≤10 moderate or severe migraine attacks per month in each of the two months prior to Screening (Visit 1).
4. Meet the following requirements:

   1. Is a male who agrees to all of the following:

      * If partner is a non-pregnant female of childbearing potential: To use an appropriate method of contraception, including a condom with spermicidal cream or jelly, from the first dose of study drug until ≥72 hours after the last dose of study drug (i.e. Period 3). A male participant who has had a vasectomy procedure must use a condom but is not required to use spermicidal cream or jelly.
      * If partner is pregnant: To use a condom from the first dose of study drug until ≥72 hours after the last dose of study drug.

      Note: Contraception/condom requirements are waived if partner is NOT of childbearing potential (i.e. is male or is a female who is post-menopausal or surgically sterile [post-hysterectomy or bilateral salpingectomy]).
      * To not donate sperm from the first dose of study drug until ≥ 72 hours after the last dose of study drug.

      OR
   2. Is a female who is of non-childbearing potential defined by at least 1 of the following criteria:

      * Postmenopausal defined as one of the following: a minimum of 12 months of spontaneous amenorrhea OR a minimum of 6 months of spontaneous amenorrhea with a Screening serum follicle-stimulating hormone (FSH) level >40 mIU/mL OR at least 6 weeks post-bilateral oophorectomy (with or without hysterectomy).
      * Post hysterectomy or bilateral salpingectomy, based on the participant's recall of their medical history.
      * If pre-menopausal, they must agree to not donate eggs from the first dose of study drug until 30 days after the last dose study drug.

   OR c. Is a female of reproductive potential and:
   * agrees to not donate eggs from the first dose of study drug until 30 days after the last dose study drug.

   AND
   * agrees to remain abstinent from heterosexual activity*,** or
   * agrees to use (or have their partner use) a birth control method that is highly effective**. Acceptable methods of birth control are:

     * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation
     * Progestogen-only contraception (e.g. oral, injectable, implant) associated with inhibition of ovulation
     * Intrauterine device (IUD)
     * Intrauterine hormone-releasing system (IUS)
     * Bilateral tubal occlusion
     * Vasectomized partner * Abstinence can be used as the sole method of contraception if it is in line with the participant's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and ethics committees. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception.

       * Note: Participants must agree that they will not attempt to become pregnant during the cycles of study drug administration or the menstrual cycle following the last dose of study medication.
5. Voluntarily agrees to participate in the study by giving written informed consent.
6. Is able to read, understand, and complete the study questionnaires and diary.
7. Be willing and able to comply with the study schedule of visits and all trial procedures and restrictions.
8. Be willing to use their own personal, qualified smartphone to download study-specific eDiary applications for use during the study.

KEY EXCLUSION CRITERIA:

1. Is a female who is pregnant, breast-feeding or intends to become pregnant during the planned course of the study. Note: Female participants of childbearing potential must have a negative serum pregnancy test (beta-human chorionic gonadotropin [beta-hCG]) performed by the central laboratory prior to enrollment in the study and negative urine pregnancy result at the randomization visit.

   Migraine history-related exclusion criteria
2. Has difficulty distinguishing his/her migraine attacks from tension-type headaches.
3. Has a history of predominantly mild migraine attacks or migraines that usually resolve spontaneously in less than two hours.
4. Has more than 15 headache-days per month or has taken medication for acute headache on more than 10 days per month in any of the three months prior to Screening (Visit 1).
5. Has brainstem (also known as [a.k.a.] basilar-type) or hemiplegic migraine headache, or retinal migraine.
6. Was >50 years old at age of first migraine onset.
7. Is taking migraine prophylactic medication where the prescribed daily dose has changed during the 3 months prior to Screening (Visit 1) or anticipates any change during the study.
8. Stopped preventive migraine medication(s) within 30 days prior to Screening for small molecules or 90 days for antibodies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2025-08-12 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with pain freedom | 2 hours post-dose

SECONDARY OUTCOMES:
Percentage of participants with freedom from the most bothersome symptom | 2 hours post-dose
Percentage of participants who report pain relief | 2 hours post-dose
Percentage of participants who experienced 1 or more treatment-emergent adverse events (AEs) | up to 7 days after the last dose of study medication
Percentage of participants who experienced 1 or more treatment-emergent serious adverse events (SAEs) | up to 7 days after the last dose of study medication

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Excell Research, Inc., Oceanside, California
  - DelRicht Research - Atlanta, Atlanta, Georgia
  - Clinical Research Atlanta - Stockbridge, Stockbridge, Georgia
  - Chicago Headache Center and Research Institute, Chicago, Illinois
  - Collective Medical Research, Overland Park, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - DelRicht Research - Prairieville, Prairieville, Louisiana
  - Clinical Research Institute, Minneapolis, Minnesota
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Dent Neurosciences Research Center, Amherst, New York
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Headache Wellness Center, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - DM Clinical Research - Bellaire, Houston, Texas
  - APD Clinical Research, Splendora, Texas
  - Health Research of Hampton Roads, Inc., Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No